CLINICAL TRIAL: NCT03139734
Title: Sacral Neuromodulation for Pelvic Pain Associated With Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seinajoki Central Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other); Oulu University Hospital (Other); Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Adrian Zegrea, MD, Principal Investigator, Seinajoki Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDONEMO
Record Dates: First submitted 2017-04-07; First posted 2017-05-04 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Endometriosis
Keywords: Sacral Nerve Modulation
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacral neuromodulation (Other): The purpose of this study is to find out if Sacral Neuromodulation is an effective treatment for pelvic pain associated with endometriosis.
  Interventions: Device: Sacral Neuromodulation

INTERVENTIONS:
Device: Sacral Neuromodulation — S3 nerve root (sometimes S4) is stimulated with low electrical current via an electrode placed through a sacral foramen. This electrode is connected to a stimulator resembling a cardiac pacemaker.
  Other Names: Sacral Nerve Stimulation; Sacral Nerve Modulation

SUMMARY:
The purpose of this study is to find out if sacral neuromodulation is an effective treatment for pelvic pain associated with surgically treated endometriosis.

DETAILED DESCRIPTION:
Endometriosis is typically associated with severe pelvic pain and pain is often combined with dysfunctional symptoms of the urinary bladder and the bowel. Endometriosis impairs the health-related quality of life and pain is the main reason for the decreased quality of life. When the primary endometriosis treatments, i.e. hormonal therapy and surgery, fail to alleviate pain or symptoms recur after successful treatment, the options are often limited. Recurrent or long-lasting endometriosis pain commonly involves neuropathic pain component with periferal or central sensitisation to pain. This kind of pain is likely more resistant to traditional endometriosis treatments and thus neuromodulation offers a logical treatment option.

There are some case series and at least one randomized trial describing the effect of Sacral Neuromodulation in chronic pelvic pain associated with interstitial cystitis and painful bladder syndrome. These reports indicate that Sacral Neuromodulation may be effective in treating chronic pelvic pain but the level of evidence is low. There is one report on long-term pelvic pain with Visual Analogue Scale score dropping from 8.1 to 2.1 and the effect lasting for five years. There are also few case reports on different difficult sacral area pain conditions treated successfully with Sacral Nerve Modulation. The common consensus seems to be that further studies are needed on the effects of Sacral Neuromodulation on chronic pelvic pain.

This study aims to evaluate if sacral neuromodulation alleviates pelvic pain symptoms and related dysfunctional symptoms in surgically treated endometriosis patients and improves their health-related quality of life. The treating gynecologist does the screening for suitable patients and a signed informed consent is needed from the patients prior to entering the study. A test pulse generator is placed uni- or bilaterally under local or general anesthesia and used during a 2-3-week test period. A permanent pulse generator is placed if marked improvement of symptoms is detected, the patient is satisfied with the treatment and willing to continue. Women not responding to sacral neuromodulation will not receive a permanent generator. They are asked to continue in the 3 year follow-up and they serve as the control group if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Life interfering pelvic pain with no other obvious pathology than endometriosis, that has been histologically confirmed at previous surgery.
* History of radical or fertility sparing endometriosis surgery either without obvious recurrent or residual endometriosis at gynecological examination and pelvic imaging (transvaginal ultrasound examination and/or pelvic MRI) or with recurrent or residual endometriosis, but re-operation is not desirable.
* Other treatment options, i.e. hormonal treatments and pain medications, are in use or have been tested, but they are ineffective or not possible to use due to contraindications or side effects..

Exclusion Criteria:

* Present or future desire to become pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — gender identity
Enrollment: 50 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain intensity and frequency | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  Pain is evaluated with Patient's pain diary: self-reported daily pain intensity (NRS 0-10) for dysmenorrhea, non-cyclic pelvic pain, dyschezia, dysuria and dyspareunia during one month period. NRS= numerical rating scale with 0 meaning "no pain" and 10 meaning "Worst pain one can imagine"

SECONDARY OUTCOMES:
Pelvic pain intensity | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  Pain is evaluated with Brief Pain Inventory Questionnaire at clinical visits
Disease specific health-related quality of life | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  Endometriosis Health Profile Questionnaire (EHP-30)
General health-related Quality of life | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  15D-measure
Sexual health-related quality of life | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  McCoy Female Sexuality Questionaire
Pelvic organ dysfunction symptoms | Change measures at baseline, before and during Sacral neuromodulation test period and 1-2 months after initiation of the modulation and then every 6 months for 3 years
  Pelvic Floor Distress Inventory (PFDI-20)
Patient satisfaction with sacral neuromodulation treatment | Change measures 1-2 months after initiation of the sacral neuromodulation and then every 6 months for 3 years
  Evaluation of satisfaction with sacral neuromodulation treatment evaluated with NRS 0-10 (0= totally dissatisfied and 10= totally satisfied)

OTHER OUTCOMES:
The need for sick-leave due to pelvic pain/endometriosis | Change measures: retrospectively asked at baseline and then every 6 months during the 3 year follow-up
  Number of sick-leave days/week during 6 months period

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo Tammela, Principal Investigator — Tampere University Hospital
Locations (1):
- Turku University Hospital (Tyks) Main Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No